CLINICAL TRIAL: NCT04026906
Title: Skin Glue to Reduce Peripheral Intravenous Catheter Failure Rate in Children: A Randomized Controlled Trial
Brief Title: Skin Glue to Reduce Intravenous Catheter Failure in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Maala Bhatt, Pediatric Emergency Medicine Staff Physician, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19/09E
Record Dates: First submitted 2019-07-11; First posted 2019-07-19 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Dislodged Catheter
Keywords: skin glue; dermabond; randomized controlled trial; intravenous catheter

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Skin Glue (Experimental): Patients in the intervention group will receive standard peripheral intravenous catheter (PIVC) securement (with cloth-bordered transparent polyurethane dressing (Tegaderm® I.V. Advanced) and tape). In addition they will receive a drop of cyanoacrylate glue (Dermabond® topical skin adhesive) at both the PIVC insertion site and under the hub of the catheter.
  Interventions: Device: Cyanoacrylate glue
- Standard Care (Placebo Comparator): Patients in the control group will receive standard PIVC placement with cloth-bordered transparent polyurethane dressing (Tegaderm® I.V. Advanced) and tape.
  Interventions: Other: Transparent polyurethane dressing

INTERVENTIONS:
Device: Cyanoacrylate glue — One drop of cyanoacrylate glue will be applied to the intravenous (IV) insertion site and another drop under the hub of the IV catheter
  Arms: Skin Glue
Other: Transparent polyurethane dressing — The IV will be secured in the usual manner with tape and a transparent dressing.
  Arms: Standard Care

SUMMARY:
Intravenous (IV) catheter placement is the most common medical procedure in emergency department settings. IVs are used to deliver medications, fluids and blood products to patients. At the Children's Hospital of Eastern Ontario, approximately three-quarters of children admitted to hospital have an IV inserted while they are in the emergency department. However, a challenge associated with IVs is that they sometimes stop working or fall out before treatment has been completed (this is known as IV failure). When IVs fail, a new IV often needs to be placed. Children rank IV placement as one of the leading causes of pain in the hospital setting. The investigators are interested in understanding whether there are strategies that can help keep IVs in place longer for children admitted to hospital.

Previous studies investigating whether certain types of bandages over IV sites are helpful in keeping IVs in longer found all bandages performed about the same. However, a recent study of adult patients showed that using medical-grade skin glue to secure the IV significantly reduced IV failure rates when compared to usual care. There have been no similar studies in children. The objective of this study is to understand whether placement of skin glue at IV insertion sites is effective in decreasing IV failure rates in children. This study will take place in the emergency department at Children's Hospital of Eastern Ontario (CHEO). Consenting children will be randomly assigned to receive IV placement either with or without skin glue (one drop at the IV insertion site and another drop under the hub of the catheter), along with otherwise standard securement with a transparent dressing. The investigators will look at the numbers of children in each group whose IVs fail before their intended treatment course is complete. This study has the potential to improve patient and family satisfaction, decrease nursing workload and reduce healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

1. Age 0 days to 18 years
2. Patient must require a PIVC as part of their management plan
3. Patient must be physically in the ED at the time of PIVC insertion

Exclusion Criteria:

1. At the time of insertion, the treating physician anticipates the patient will likely be discharged from the ED (with or without the PIVC in place)
2. Known allergy to skin glue, glue removal wipe, or standard catheter securement materials
3. Active infection at site of PIVC insertion
4. Insurmountable language barrier (patient's parent/guardian is unable to understand English or French well enough to give informed consent and participate in follow-up)
5. Previous enrolment in the trial
6. PIVC is expected to be used for chemotherapy (note: these are changed every 4 days even with good blood return)
7. Life-threatening or critical presentation in which consent is unable to be obtained

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 557 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
PIVC failure before the intended intravenous treatment course is complete. | Measured at the point at which the PIVC fails, up to 14 days
  PIVC failure is defined by a composite of dislodgement, occlusion, signs of infection, and phlebitis. Dislodgement is defined as subcutaneous extravasation, accidental removal by patient or staff, or history that the PIVC "fell out". Occlusion is defined as an inability to flush the catheter with 2-3ccs of normal saline or history that the PIVC was "not working". Infection is defined as presence of pus, erythema, pain, and/or swelling around the PIVC site in keeping with a clinical suspicion of infection or cellulitis. Phlebitis is defined as a painful, palpable, cord-like vein.If the PIVC fails (as per the above definition) before an order is written to discontinue the PIVC, it will be determined the device failed before the treatment course was complete.

SECONDARY OUTCOMES:
Time to PIVC failure | Time from PIVC insertion to either a) PIVC failure or b) when PIVC is not longer needed for treatment, up to 14 days
  Time from PIVC insertion to failure (measured in hours)
PIVC failure or removal as a result of each of the following: a) dislodgement, b) occlusion, c) infection, and d) phlebitis | End of study period, up to 14 days
  Numerator: number of PIVCs that fail; Denominator: Total number of PIVCs inserted
Pain on PIVC removal as experienced by the patient or observed by the caregiver | Measured at the time of PIVC removal, up to 14 days
  Measured using the Visual Analogue Scale
Difficulty of PIVC removal | Measured at the time of PIVC removal, up to 14 days
  measured by the bedside nurse using a 4-point Likert scale

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Of Eastern Ontario, Ottawa, Ontario, Canada